CLINICAL TRIAL: NCT00856232
Title: Oxygen Therapy for the Treatment of Undifferentiated Headache in the Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Responsible Party: Principal Investigator, rwjms-ed, Assistant Professor, Rutgers, The State University of New Jersey
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0220080056
Record Dates: First submitted 2009-03-04; First posted 2009-03-05 (Estimated); Results first posted 2013-05-03 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-03

CONDITIONS: Headache
Keywords: Headache; Cephalgia; Migraine
MeSH Terms: conditions — Headache; Migraine Disorders | interventions — Air; Oxygen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard therapy (No Intervention): Standard emergency department evaluation and treatment for headache
- Medical Air (Placebo Comparator): Air inhalation at 15L / min x 15 minutes followed by standard emergency department evaluation and treatment for headache
  Interventions: Biological: Medical Air
- Oxygen (Experimental): Oxygen inhalation at 15 L/min for 15 minutes followed by standard emergency department evaluation and treatment for headache
  Interventions: Biological: Oxygen

INTERVENTIONS:
Biological: Medical Air — Compressed medical air
  Arms: Medical Air
Biological: Oxygen — Medical Oxygen
  Arms: Oxygen

SUMMARY:
This study will randomly assign emergency department patients seeking treatment for a headache to one of three groups. The first group will receive standard emergency care as determined by the treating physician, the second group will breathe high flow air by facemask for 15 minutes, and the third group will breathe high flow oxygen by face mask for 15 minutes. The patients will be questioned in the beginning of their treatment and at 2, 5, 10, 15 and 30 minutes after it's begun about the intensity of their headache and how much relief they are experiencing from their treatment. Concentration of carbon dioxide exhaled by patients will also be recorded at 0, 2, 5, 10, 15 and 30 minutes. After fifteen minutes, the patients in groups 2 and 3 will continue with standard emergency care, which can include any treatment their physician sees fit. Patients in all three groups will receive a stopwatch in the beginning of their emergency department visit and record the total extent of time their headache will take to resolve.

DETAILED DESCRIPTION:
Thorough description provided in brief summary.

ELIGIBILITY:
Inclusion Criteria:

* All patients who describe a painful sensation in the head as one of the primary reasons for their visit to the ED.

Exclusion Criteria:

* patients who need immediate oxygen after triage: Recent fire or carbon monoxide exposure_______ O2 saturation 94% or less on room air on triage vitals ______ patient arrives on supplemental oxygen_______ patient reports shortness of breath_______
* patients in whom 100% oxygen is contraindicated, potentially undesirable, or controversial: history of COPD_______ possible cardiac ischemia (mouth / jaw / neck / shoulder / chest / abdomen pain or pressure)_______ possible stroke (new focal weakness or numbness, speech, hearing or vision deficit, bowel or bladder incontinence or retention)_____
* patients unable to tolerate the gas treatment: patient not able to tolerate a face mask_______ patient requests immediate treatment with another preferred therapeutic agent_______
* treating physician or nurse request to discontinue the study at any point_______
* patients who have diminished decision-making capacity history of mental retardation or pervasive developmental disorder_______ patient not awake and alert_______ patient not oriented to self, month and year, and current location_______ patient unwilling or unable to fully participate in the research associate interview and consent process_______
* patients who are at risk for intracranial hemorrhage history of intracranial aneurythm, hemorrhage, surgery, or tumor_______ current headache began after trauma_______ current headache began after using elicit drugs_______
* patients who are at high risk for intracranial infection fever > 100.4 F on triage vitals_______ complaining of recent onset neck stiffness_______
* patients who are at high risk for extracranial head pathology ear pain or drainage_______ tooth or gum pain_______ headache localized to a skin lesion on the head______
* patient is potentially critically ill active bleeding from any source_______ heart rate <60 or >130 on triage vitals_______ systolic blood pressure <90 or >180 on triage vitals_______ respiratory rate < 10 or >30 on triage vitals_______
* patient is younger than 21_______
* patients who know or suspect they are pregnant _____

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2009-01; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boris D Veysman, M.D., Principal Investigator — Department of Emergency Medicine, UMDNJ - Robert Wood Johnson Medical School
Locations (1):
- Robert Wood Johnson University Hospital Emergency Department, New Brunswick, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Air at 15L/Min: Air inhalation at 15L / min x 15 minutes followed by standard emergency department evaluation and treatment for headache
Period: Overall Study
Arm/Group | Standard Therapy | Air at 15L/Min | Oxygen
Started | 26 | 29 | 36
Completed | 26 | 29 | 36
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Therapy | Air at 15L/Min | Oxygen | Total
Number analyzed (Participants) | 26 | 29 | 36 | 91
Age, Categorical [Number; unit: participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | NA — Age data not collected as part of IRB protocol | NA — Age data not collected as part of IRB protocol | NA — Age data not collected as part of IRB protocol | NA — Total not calculated because data are not available (NA) in one or more arms.
  >=65 years | NA — Age data not collected as part of IRB protocol | NA — Age data not collected as part of IRB protocol | NA — Age data not collected as part of IRB protocol | NA — Total not calculated because data are not available (NA) in one or more arms.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | NA — gender data not collected as part of IRB protocol | NA — gender data not collected as part of IRB protocol | NA — gender data not collected as part of IRB protocol | NA — Total not calculated because data are not available (NA) in one or more arms.
  Male | NA — gender data not collected as part of IRB protocol | NA — gender data not collected as part of IRB protocol | NA — gender data not collected as part of IRB protocol | NA — Total not calculated because data are not available (NA) in one or more arms.
Region of Enrollment [Number; unit: participants]
  United States | 26 | 29 | 36 | 91

OUTCOME MEASURES:

1. Secondary Outcome: Length of Stay in the Emergency Department(Min)
Description: Length of stay was reported as time elapsed in minutes from subject's arrival as a patient to the Emergency Department to patient's discharge from the Emergency Department.
Time Frame: Study duration
Measure: Mean (Standard Deviation); unit: Minutes
Groups:
- Medical Air at 15L/Min: Air inhalation at 15L / min x 15 minutes followed by standard emergency department evaluation and treatment for headache
- Oxygen at 15 L / Min: Oxygen inhalation at 15 L/min for 15 minutes followed by standard emergency department evaluation and treatment for headache
Arm/Group | Standard Therapy | Medical Air at 15L/Min | Oxygen at 15 L / Min
Number analyzed (Participants) | 26 | 29 | 36
Minutes | 177.5 (109) | 210.7 (134.9) | 118.7 (145.8)

2. Primary Outcome: Time to Relief (Min)
Description: Time to relief is a measure of time reported by a stopwatch the patients were provided in the beginning of the study, which showed elapsed time in minutes for patients to perceive that they no longer had a headache.
Time Frame: study duration
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Standard Therapy | Air at 15L/Min | Oxygen
Number analyzed (Participants) | 26 | 29 | 36
Minutes | 92.2 (84.4) | 83.9 (45.3) | 35.4 (29.8)

ADVERSE EVENTS:
Arm/Group | Standard Therapy | Air at 15L/Min | Oxygen
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/29 | 0/36
Other Adverse Events (participants affected / at risk) | 0/26 | 0/29 | 0/36

LIMITATIONS AND CAVEATS:
Limited number of subjects due to difficulty with recruitment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No